CLINICAL TRIAL: NCT06142760
Title: Daily AI-based Treatment Adaptation Under Weekly Offline MR-guidance in Chemoradiotherapy for Cervical Cancer 1 AIM-C1
Brief Title: MR-guidance in Chemoradiotherapy for Cervical Cancer
Acronym: AIM-C1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juergen Debus (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, Department head, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-AIM-C1
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MR-guided radiation — Dayly artifical intelligence-based treatment adaptation under weekly offline MR-guidance

SUMMARY:
Concurrent chemoradiotherapy (CCRT), consisting of external beam radiotherapy (EBRT) and chemotherapy, followed by brachytherapy (BT) is the standard of care for patients with locally advanced cervical carcinoma. In current clinical practice, conventionally, one radiotherapy plan based on the initial planning computed tomography (CT) and magnetic resonance imaging (MRI) scan of the pelvis is applied for the complete 5-6 weeks of EBRT. However, there is a high degree of cervix and uterus motion in the pelvis due to different fillings of the bladder and the bowel. Consequently, large safety margins are required to compensate for organ movement, potentially leading to higher toxicity. Lately, daily high-quality cone-beam CT (CBCT) guided adaptive radiotherapy, aided by artificial intelligence (AI), became clinically available. Due to the improved soft-tissue contrast, the treatment plan can now be online adapted to the current position of the tumor and the adjacent organs-at-risk (OAR), while the patient is lying on the treatment couch. Moreover, the German Research Cancer Center offers the unique possibility of additional weekly magnetic resonance imaging (MRI) in treatment position using a shuttle system. Daily CBCT-adapted EBRT in combination with weekly MRI in treatment position might therefore offer superior sparing of surrounding OAR and consequently reduction of treatment-associated side-effects.

However, to the investigators knowledge, no toxicity data for daily CBCT/AI adaptive EBRT of locally advanced cervical cancer with additional MR-guidance exists. The AIM-C1 trial therefore aims to assess the potential of daily CBCT adaptive and AI aided EBRT combined with additional weekly offline MR-guidance in treatment position using a shuttle system.

DETAILED DESCRIPTION:
This trial will be conducted as a prospective, one-armed phase II study in 40 patients with cervical carcinoma (FIGO stage IB, IIA, IIB, IIIA, IIIB, IIIC1), age ≥ 18 years, Karnofsky Performance Score ≥ 70%. CCRT will consist of 50.4Gy external beam radiotherapy (EBRT) with concurrent cisplatin 40mg/m² as standard of care in Germany, followed by 27Gy of BT in 4 fractions of 7Gy.

The primary endpoint of the trial will be the occurrence of overall early bowel and bladder toxicity CTCAE grade 2 or higher assessed within the first 3 months with NCI CTCAE Version 5.0.

Secondary outcomes to be investigated are clinical feasibility of daily CBCT-guided and weekly MR-guided plan adaptation, local tumor control, distant tumor control, progression-free survival, overall survival, quality of life, acquisition and comparison of different MRI sequences, technical analyses of treatment, adaptation frequency and morphological as well as functional tumor characteristics of the MRI.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven cervical cancer including squamous-cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma
* FIGO stage IB, IIA, IIB, IIIA, IIIB, IIIC1
* indication and eligibility for definitive chemoradiotherapy including brachytherapy discussed in an interdisciplinary tumor board
* Karnofsky performance score ≥ 70%
* 18-80 years of age
* Capacity of the patient to consent to participation in the study

Exclusion Criteria:

* FIGO stage IIIC2 and IV
* Paraaortic lymphatic node metastases
* small cell neuroendocrine cancer, melanoma and other rare cancers of the cervix
* previous radiotherapy of the pelvic region
* previous total or partial hysterectomy
* neoadjuvant chemotherapy
* contraindications against performing contrast-enhanced MRI scans (pacemakers, other implants making MRI impossible, allergy to gadolinium (GD)-based contrast agent)
* claustrophobia
* pregnant or lactating women
* other primary malignancies within 5 years before except carcinoma in situ of the cervix and basal cell carcinoma of the skin
* patient is enrolled in another study, that could influence the outcome of the presented study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-related bladder toxicity | within 3 month after completion of radiation treatment
  Occurrence of bladder toxicity grade 2 or higher according to CTCAE V5.0
Treatment-related bowl toxicity | within 3 month after completion of radiation treatment
  Occurrence of bowl toxicity grade 2 or higher according to CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No